CLINICAL TRIAL: NCT03892564
Title: A 4-Day, Randomized Study to Evaluate the Potential of MC2-01 Cream to Induce a Phototoxicity Skin Reaction in Healthy Subjects, Using a Controlled Photopatch Test Design
Brief Title: Evaluation of Potential Phototoxicity Skin Reaction After Use of MC2-01 Cream
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MC2 Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MC2-01-C9
Record Dates: First submitted 2019-03-20; First posted 2019-03-27 (Actual); Results first posted 2020-02-12 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Phototoxicity
MeSH Terms: conditions — Dermatitis, Phototoxic | interventions — Radiation

STUDY DESIGN:
Intervention Model Description: One treatment with MC2-01 Cream, MC2-01 vehicle and control on defined applications site (N=5), followed by irradiation/non-irradiation and evaluation 24 or 48 hours post irradiation, within subject comparison model
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- MC2-01 Cream, irradiation (Experimental): One applications with MC2-01 Cream (calcipotriene/betamethasone dipropionate, w/w 0.005%/0.064%) cream, followed by irradiation
  Interventions: Drug: MC2-01 Cream, irradiation
- MC2-01 Cream, no irradiation (Experimental): One application of MC2-01 Cream (CAL/BDP, 0.005%/0.064%), no irradiation. Visual evaluation of application site using a visual scale that rated the degree of erythema, edema and other signs of cutaneous irritation
  Interventions: Drug: MC2-01 Cream, no irradiation
- MC2-01 vehicle, irradiation (Experimental): One application of MC2-01 vehicle, followed by irradiation. Visual evaluation of application site using a visual scale that rated the degree of erythema, edema and other signs of cutaneous irritation
  Interventions: Drug: MC2-01 vehicle, irradiation
- MC2-01 vehicle, no irradiation (Experimental): One application of MC2-01 vehicle, no irradiation. Visual evaluation of application site using a visual scale that rated the degree of erythema, edema and other signs of cutaneous irritation
  Interventions: Drug: MC2-01 vehicle, no irradiation
- Control, irradiation (Experimental): Untreated, irradiated site. Visual evaluation of application site using a visual scale that rated the degree of erythema, edema and other signs of cutaneous irritation
  Interventions: Drug: Control, irradiation

INTERVENTIONS:
Drug: MC2-01 Cream, irradiation — One application of MC2-01 Cream, followed by irradiation. Visual evaluation of application site using a visual scale that rated the degree of erythema, edema and other signs of cutaneous irritation
  Arms: MC2-01 Cream, irradiation
Drug: MC2-01 Cream, no irradiation — One application of MC2-01 Cream. Visual evaluation of application site using a visual scale that rated the degree of erythema, edema and other signs of cutaneous irritation
  Arms: MC2-01 Cream, no irradiation
Drug: MC2-01 vehicle, irradiation — One application of MC2-01 vehicle, followed by irradiation. Visual evaluation of application site using a visual scale that rated the degree of erythema, edema and other signs of cutaneous irritation
  Arms: MC2-01 vehicle, irradiation
Drug: MC2-01 vehicle, no irradiation — One application of MC2-01 vehicle. Visual evaluation of application site using a visual scale that rated the degree of erythema, edema and other signs of cutaneous irritation
  Arms: MC2-01 vehicle, no irradiation
Drug: Control, irradiation — Untreated, irradiated site. Visual evaluation of application site using a visual scale that rated the degree of erythema, edema and other signs of cutaneous irritation
  Arms: Control, irradiation

SUMMARY:
This trial is a 4-day, randomized study to determine the phototoxic potential of MC2-01 Cream when topical application to healthy skin is followed by light exposure.

DETAILED DESCRIPTION:
This study evaluates the potential of MC2-01 (CAL/BDP 0.005/0.042w/w%) Cream to cause a phototoxic reaction using a controlled photopatch test design. Because MC2-01 Cream is formulated for topical use and have shown to absorb light, it is necessary to determine the potential of this product to cause a phototoxic reaction after topical application and irradiation of the skin.

ELIGIBILITY:
Inclusion Criteria:

* Is a healthy male or female
* Is 18 years of age or older
* Agree not to participate in any clinical or patch test studies at Day 1 through study completion
* Females of childbearing potential must use a highly effective method of contraception for one month prior to Screening and until the end of study visit has been performed
* in the case of a female of childbearing potential, has a negative urine pregnancy test on Day 1 prior to randomization and are willing to submit to a urine pregnancy test at the end of study
* In the case of a female of non-childbearing potential, has had a hysterectomy or is postmenopausal
* Is free of any systemic or dermatological disorder, which, in the opinion of the Investigator, will interfere with the study results or increase the risk of AEs.
* Has uniformly-colored skin on the intrascapular region of the back which will allow discernment of erythema, and has Fitzpatrick skin types I, II or III
* Complete a medical screening procedure
* Read, understand and sign an informed consent

Exclusion Criteria:

* Has a history of photosensitivity or photoallergy
* Has any visible skin disease at the application site which, in the opinion of the Investigator, will interfere with the evaluation of the test site reaction
* Current or past history of hypercalcemia, vitamin D toxicity, severe renal insufficiency or severe hepatic disorders
* Is using systemic/topical corticosteroids within 3 weeks prior to and/or during the study or systemic/topical antihistamines 72 hours prior to and during the study
* Is not willing to refrain from using systemic/topical anti-inflammatory analgesics (81 mg aspirin and occasional use of acetaminophen will be permitted)
* Are taking medication known to cause phototoxic reaction
* Is using medication which, in the opinion of the Investigator, will interfere with the study results
* Is unwilling or unable to refrain from the use of sunscreens, cosmetics, creams, ointments, lotions or similar products on the back during the study
* Has psoriasis and/or atopic dermatitis/eczema
* Has a known sensitivity or allergy to constituents of the materials being evaluated
* Is a female who is pregnant, plans to become pregnant during the study, or is breast feeding a child
* Has damaged skin in or around the test sites, including sunburn, excessively deep tans, uneven skin tones, tattoos, scars excessive hair, numerous freckles or other disfigurations of the test site
* Has received treatment for any type of internal cancer within 5 years prior to study entry
* Has a history of, or are currently being treated for skin cancer and/or hepatitis
* Has a history or, or is currently being treated for diabetes
* Has any condition that might compromise study results
* Is expected to sunbathe or use tanning salons during the study
* Has a history of adverse response to UV-sun lamps/sunlight exposure
* Is currently participating in any clinical testing
* Has any known sensitivity to adhesives
* Has received any investigational drug(s) within 28 days from Day 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2019-02-27 (Actual); Primary Completion 2019-03-09 (Actual); Study Completion 2019-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan S Dorsik, Principal Investigator — TKL Research, Inc.
Locations (1):
- TKL Research Inc, Fair Lawn, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
Single site study

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Subject First Visit: 27-Feb-2019. Last Subject Last Visit: 09-Mar-2019
Pre-assignment Details: The study consist of a screening day + treatment period of 4 consecutive days.
  The study is a within-subject comparison study of MC2-01 cream and vehicle. The products were each applied to 2 sites; one was irradiated and other non-radiated. The irradiated and non-irradiated sites were compared to each other and with an untreated irradiated site.
Groups:
- Test Sites: 5 test sites on the subject's back defined as:
  1. - One application with MC2-01 Cream (calcipotriene/betamethasone dipropionate, w/w 0.005%/0.064%) cream, followed by irradiation
  2. - One application with MC2-01 Cream Calcipotriene/betamethasone dipropionate, w/w 0.005%/0.064%) cream, non-irradiation
  3. - One application of MC2-01 vehicle, followed by irradiation.
  4. - One application of MC2-01 vehicle, non-irradiation.
  5. - Control site (no application, only irradiated)
  to perform visual evaluation of application site of erythema, edema and other signs of cutaneous irritation
Period: Overall Study
Arm/Group | Test Sites
Started | 35
MC2-01 Cream + Irridiation | 35
MC2-01 Cream + Non-irridiation | 35
MC2-01 Vehicle + Irridiation | 35
MC2-01 Vehicle + Non-irridiation | 35
Control Site | 35
Completed | 33
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Test Sites
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.0 (9.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 34
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 35
Fitzpatrick Skin Type [Count of Participants; unit: Participants] — Fitzpatrick Skin Type is a method to describe the individual skin types in the following 6 categories:
  I - Pale white skin, blue/hazel eyes, blond/red hair II - Fair skin, blue eyes III - Darker white skin IV - Light brown skin V - Brown skin VI - Dark brown or black skin
  Participants
    II | 9
    III | 26

OUTCOME MEASURES:

1. Primary Outcome: Within-subject Comparison and Evaluator Rating of Possible Dermal Reactions (Erythema, Edema and Other Signs of Cutaneous Irritation), After Application of MC2-01 Cream, MC2-01 Vehicle or Untreated at Defined Test Sites, Followed by Irradiation
Description: MC2-01 Cream, MC2-01 vehicle will be applied each to two sites. One further site will function as control site and will remain untreated. 24 hours after product application, the test sites, including the untreated control site will be evaluated for cutaneous reaction. One set of MC2-01 and MC2-01 vehicle + the untreated control site will be designated for irradiation and the other set will remain non-irradiated. Possible changes in dermal reactions (erythema, edema and other signs of cutaneous irritation) at the 5 test sites, 24 and 48 hours post-irradiation is the outcome measure of the study
Time Frame: Baseline, before irradiation
Population: As the study is a within subject evaluation of dermal reactions, after application on two sites with MC2-01 cream and two sites with MC2-01 vehicle, followed by either irradiation or non-irradiation + a irradiated control site, all subjects received all 5 different treatments.
Measure: Count of Participants; unit: Participants
Groups:
- Test Sites: 1. - One application with MC2-01 Cream (calcipotriene/betamethasone dipropionate, w/w 0.005%/0.064%) cream, followed by irradiation
  2. - One application with MC2-01 Cream Calcipotriene/betamethasone dipropionate, w/w 0.005%/0.064%) cream, non-irradiation
  3. - One application of MC2-01 vehicle, followed by irradiation.
  4. - One application of MC2-01 vehicle, non-irradiation.
  5. - control, irradiated
Arm/Group | Test Sites
Number analyzed (Participants) | 33
Participants
  MC2-01 Cream, irradiation: No erythema/edema | 33
  MC2-01 Cream, irradiation: Mild, definite erythema/edema | 0
  MC2-01 Cream, non-irradiation: No erythema/edema | 33
  MC2-01 Cream, non-irradiation: Mild, definite erythema/edema | 0
  MC2-01 vehicle, irradiation: No erythema/edema | 32
  MC2-01 vehicle, irradiation: Mild, definite erythema/edema | 1
  MC2-01 vehicle, non-irradiation: No erythema/edema | 32
  MC2-01 vehicle, non-irradiation: Mild, definite erythema/edema | 1
  Control site: No erythema/edema | 33
  Control site: Mild, definite erythema/edema | 0

2. Primary Outcome: Within-subject Comparison and Evaluator Rating of Possible Dermal Reactions (Erythema, Edema and Other Signs of Cutaneous Irritation), After Application of MC2-01 Cream, MC2-01 Vehicle or Untreated at Defined Test Sites, Followed by Irradiation
Description: as for outcome 1
Time Frame: 24h post-irradiation
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Test Sites: 5 test sites on the subject's back defined as:
  1. - One application with MC2-01 Cream (calcipotriene/betamethasone dipropionate, w/w 0.005%/0.064%) cream, followed by irradiation
  2. - One application with MC2-01 Cream Calcipotriene/betamethasone dipropionate, w/w 0.005%/0.064%) cream, non-irradiation
  3. - One application of MC2-01 vehicle, followed by irradiation.
  4. - One application of MC2-01 vehicle, non-irradiation.
  5. - control, irradiated
  to perform visual evaluation of application site of erythema, edema and other signs of cutaneous irritation
Arm/Group | Test Sites
Number analyzed (Participants) | 33
Participants
  MC2-01 Cream, irradiation: No erythema/edema | 21
  MC2-01 Cream, irradiation: Mild, definite erythema/edema | 12
  MC2-01 Cream, non-irradiation: No erythema/edema | 33
  MC2-01 Cream, non-irradiation: Mild, definite erythema/edema | 0
  MC2-01 vehicle, irradiation: No erythema/edema | 21
  MC2-01 vehicle, irradiation: Mild, definite erythema/edema | 12
  MC2-01 vehicle, non-irradiation: No erythema/edema | 33
  MC2-01 vehicle, non-irradiation: Mild, definite erythema/edema | 0
  Control site: No erythema/edema | 21
  Control site: Mild, definite erythema/edema | 12

3. Primary Outcome: Within-subject Comparison and Evaluator Rating of Possible Dermal Reactions (Erythema, Edema and Other Signs of Cutaneous Irritation), After Application of MC2-01 Cream, MC2-01 Vehicle or Untreated at Defined Test Sites, Followed by Irradiation
Description: as for outcome 1
Time Frame: 48h post-irradiation
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Test Sites
Number analyzed (Participants) | 33
Participants
  MC2-01 Cream, irradiation: No erythema/edema | 25
  MC2-01 Cream, irradiation: Mild, definite erythema/edema | 8
  MC2-01 Cream, non-irradiation: No erythema/edema | 33
  MC2-01 Cream, non-irradiation: Mild, definite erythema/edema | 0
  MC2-01 vehicle, irradiation: No erythema/edema | 25
  MC2-01 vehicle, irradiation: Mild, definite erythema/edema | 8
  MC2-01 vehicle, non-irradiation: No erythema/edema | 33
  MC2-01 vehicle, non-irradiation: Mild, definite erythema/edema | 0
  Control site: No erythema/edema | 25
  Control site: Mild, definite erythema/edema | 8

ADVERSE EVENTS:
Time Frame: AEs were collected/assessed from the time of the informed consent form was signed by the subject at the screening visit and during the test phase, which consisted of in total of 4 days. the 4th day was considered the last visit for the subjects. AEs assessed as reasonably possibly related to the trial medication had to be followed until they were resolved or until the medical condition of the subject was stable.
Description: 35 patients participated in the study and all patients received all 5 types of treatments. Therefore data for the 'All-Cause Mortality', 'Serious Adverse Events' and 'Other Adverse Events' fields are included and assessed for all types of medication.
Groups:
- MC2-01 Cream, Irradiation: 5 test sites on the subject's back defined as:
  1. - One application with MC2-01 Cream (calcipotriene/betamethasone dipropionate, w/w 0.005%/0.064%) cream, followed by irradiation
  2. - One application with MC2-01 Cream Calcipotriene/betamethasone dipropionate, w/w 0.005%/0.064%) cream, non-irradiation
  3. - One application of MC2-01 vehicle, followed by irradiation.
  4. - One application of MC2-01 vehicle, non-irradiation.
  5. - control, irradiated
Arm/Group | MC2-01 Cream, Irradiation
All-Cause Mortality (participants affected / at risk) | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35
Other Adverse Events (participants affected / at risk) | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-01-10): https://cdn.clinicaltrials.gov/large-docs/64/NCT03892564/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-11): https://cdn.clinicaltrials.gov/large-docs/64/NCT03892564/SAP_001.pdf